CLINICAL TRIAL: NCT03002233
Title: A Phase 1 Study to Observe Safety and Tolerability of Single and Multiple Doses of TRK-820 in Subjects on Hemodialysis and to Observe the Effect on Uremic Pruritus
Brief Title: TRK-820 Study in Subjects on Hemodialysis With or Without Uremic Pruritus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Toray Industries, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EU820UPC01
Record Dates: First submitted 2016-12-13; First posted 2016-12-23 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Uremic Pruritus
Keywords: TRK-820; Hemodialysis; Uremic Pruritus
MeSH Terms: interventions — TRK 820

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TRK-820 (Experimental): PartA: 5 μg PartB: 2.5-10 μg
  Interventions: Drug: TRK-820

INTERVENTIONS:
Drug: TRK-820
  Other Names: Nalfurafine Hydrochloride

SUMMARY:
This study is a 2-part study.

Part A is a single-dose, open-label study design to determine the PK, safety and tolerability of 5 μg TRK-820 oral administration in subjects with end-stage renal disease (ESRD) who require hemodialysis.

Part B is a multiple dose, open-label study design to determine the PK, PD, safety and tolerability of multiple doses in subjects with ESRD who require hemodialysis with refractory uremic pruritus (UP). Each subject will receive 3 doses of TRK-820 (2.5, 5 and 10 μg).

ELIGIBILITY:
Inclusion Criteria:

* Adult non-smoking male and female subjects (≥ 18 years of age) who have ESRD requiring hemodialysis, at least 3 times a week.
* Subjects has a clinical diagnosis of UP, which is uncontrolled by current medications or treatments.(Part B only)

Exclusion Criteria:

* Subject has a known hypersensitivity to opioids or the ingredients of the study medication.
* Subject has pruritus other than related to ESRD (i.e., UP).(Part B only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters: area under the time curve from time zero to 24 hours postdose(AUC0-24h) | Part A; predose to 24 hours postdose, Part B; predose to 24 hours postdose each dose
Pharmacokinetic parameters: area under the time curve from time zero to the last quantifiable concentration(AUC0-last) | Part A; predose to 60 hours postdose, Part B; predose to 48 hours postdose each dose
Pharmacokinetic parameters: area under the time curve from time zero extrapolated to infinity(AUC0-inf) | Part A; predose to 60 hours postdose, Part B; predose to 48 hours postdose each dose
Pharmacokinetic parameters: maximum observed plasma concentration (Cmax) | Part A; predose to 60 hours postdose, Part B; predose to 48 hours postdose each dose
Pharmacokinetic parameters: time to maximum plasma concentration(Tmax) | Part A; predose to 60 hours postdose, Part B; predose to 48 hours postdose each dose
Pharmacokinetic parameters: apparent elimination half-life in plasma(t½) | Part A; predose to 60 hours postdose, Part B; predose to 48 hours postdose each dose
Pharmacokinetic parameters: plasma concentration at 24 hours postdose(C24h) | Part A; 24 hours postdose, Part B; 24 hours postdose each dose
Pharmacokinetic parameters: apparent total clearance(CL/F) | Part A; predose to 60 hours postdose, Part B; predose to 48 hours postdose each dose
Pharmacokinetic parameters: terminal elimination rate(λz) | Part A; predose to 60 hours postdose, Part B; predose to 48 hours postdose each dose
Pharmacokinetic parameters: apparent distribution volume(Vz/F) | Part A; predose to 60 hours postdose, Part B; predose to 48 hours postdose each dose
Pharmacokinetic parameters: mean residence time(MRT) | Part A; predose to 60 hours postdose, Part B; predose to 48 hours postdose each dose
Pharmacodynamic parameters: Visual Analogue Scale (VAS) reduction from baseline | Part B only; Baseline to week 5

CONTACTS AND LOCATIONS:
Locations (2):
- Bulgaria, Bulgaria, Bulgaria
- Germany, Germany, Germany